CLINICAL TRIAL: NCT03280797
Title: Feasibility of a Cytokine Expression Profile in Immune Cells as an Orientation Tool in Therapeutic Decisions for Auto-inflammatory and Auto-immune Diseases
Acronym: IL-MAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: LOCAL/2016/TAT01
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other)
  Interventions: Procedure: Blood sample
- Rheumatoid arthritis patients (Other)
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — 2ml blood taken into TruCulture tube

SUMMARY:
This study will assess the feasibility of using cytokine expression profiles in blood samples as a method for evaluating rheumatoid polyarthritis

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient is at least 18 years old
* Subjects included as patients have rheumatoid polyarthritis according to ACR EULA 2010, DAS28>3.2 criteria
* Subjects included as controls are healthy volunteers who have no overexpression of cytokines

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient has had at least 3 months of specific treatment that can potentially impact cytokine profile

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Dosage of cytokines between groups | Day 0
  Concentration measured by ELISA and flow cytometry

SECONDARY OUTCOMES:
Creation of biobank | Day 0
  Storage of blood samples

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Montpellier, Montpellier
  - CHU Nimes, Nîmes